CLINICAL TRIAL: NCT05262400
Title: A PHASE 1B/2, OPEN-LABEL, MULTICENTER, DOSE ESCALATION AND DOSE EXPANSION STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, PHARMACODYNAMICS, AND ANTITUMOR ACTIVITY OF PF-07220060 IN COMBINATION WITH PF-07104091 PLUS ENDOCRINE THERAPY IN PARTICIPANTS WITH ADVANCED SOLID TUMORS
Brief Title: A Study to Learn About the Study Medicine (Called PF-07220060 in Combination With PF-07104091) In Participants With Breast Cancer and Solid Tumors
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: C4391002; 2022-002173-28 (EudraCT Number); 2023-509504-15-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2022-02-21; First posted 2022-03-02 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer; Solid Tumors
Keywords: cyclin-dependent kinase 2 (CDK2); cyclin-dependent kinase 4 (CDK4); estrogen receptor-positive/human epidermal growth factor receptor 2 negative (ER+/HER2-); estrogen receptor-positive/refractory hormone receptor positive (ER+/HER2+); hormone receptor positive/human epidermal growth factor receptor 2 negative (HR+/HER2-)
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- Part 1 Dose Escalation - Dose Level 1 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation
- Part 1 Dose Escalation - Dose Level 2 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation
- Part 1 Dose Escalation - Dose Level 3 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation
- Part 1 Dose Escalation - Dose Level 4 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation
- Part 1 Dose Escalation - Dose Level 5 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation
- Part 2A (Experimental): PF-07220060 + PF-07104091 + Fulvestrant (ER+/HER2- Breast Cancer with at least 1 prior systemic therapy for advanced or metastatic disease, including CDK4/6 inhibitor treatment and Endocrine Therapy)
  Interventions: Drug: PF-07104091 + PF-07220060 + fulvestrant dose expansion
- Part 2B (Experimental): PF-07220060 + PF-07104091 + Fulvestrant (ER+/HER2- Breast Cancer with at least 1 prior endocrine therapy and up to 1 prior line of chemotherapy for advanced or metastatic disease and no prior treatment with any CDK4/6 inhibitor for advanced disease)
  Interventions: Drug: PF-07104091 + PF-07220060 + fulvestrant dose expansion
- Part 2C (Experimental): PF-07220060 + PF-07104091 + Letrozole (ER+/HER2- Breast Cancer with no prior treatment with any CDK4/6 inhibitor for advanced disease)
  Interventions: Drug: PF-07104091 + PF-07220060 + letrozole dose expansion
- Part 1 Dose Escalation - Dose Level 6 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation
- Part 1 Dose Escalation - Dose Level 7 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation
- Part 1 Dose Escalation - Dose Level 8 (Experimental): PF-07220060 + PF-07104091 dose escalation (Breast Cancer or solid tumors)
  Interventions: Drug: PF-07220060 + PF-07104091 combination dose escalation

INTERVENTIONS:
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 1
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 2
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 3
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 4
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 5
Drug: PF-07104091 + PF-07220060 + fulvestrant dose expansion — PF-07104091 and PF-07220060 will be administered orally in combination with fulvestrant
  Arms: Part 2A
Drug: PF-07104091 + PF-07220060 + fulvestrant dose expansion — PF-07104091 and PF-07220060 will be administered orally in combination with fulvestrant
  Arms: Part 2B
Drug: PF-07104091 + PF-07220060 + letrozole dose expansion — PF-07104091 and PF-07220060 will be administered orally in combination with letrozole
  Arms: Part 2C
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 6
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 7
Drug: PF-07220060 + PF-07104091 combination dose escalation — PF-07104091 and PF-07220060 will be administered orally
  Arms: Part 1 Dose Escalation - Dose Level 8

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called PF-07220060 and PF-07104091) in people with breast cancer. This clinical study consists of 2 parts (part 1 and part 2). In part 1, we are seeking participants who:

* Have been diagnosed with Breast Cancer (BC) of either types:
* Have HR+, HER2- BC
* Refractory HR-positive/HER2-positive BC
* Have other solid tumors other than BC

In part 2, we are seeking participants who:

-Have HR-positive/HER2-negative BC Part 1 will include increasing doses of PF-07220060 with PF-07104091. In part 2, participants will take 1 of 2 study medicine combinations. This will help us decide the highest amount of study medicines that can be safety given to people. All participants in this study will receive PF-07220060 with PF-07104091 by mouth. We will compare participant experiences to help us determine if PF-07220060 with PF-07104091 is safe and effective. Participants will take part in this study for about 2 years. During this time, they will receive the study medicine, an x-ray imaging, and will be observed for safety and effects of the study medicines.

ELIGIBILITY:
Inclusion Criteria

* Part 1: Breast Cancer (BC)
* HR+, HER2- BC
* Refractory HR-positive/HER2-positive BC
* Part 1: Solid Tumors other than BC
* Part 2:
* HR-positive/HER2-negative BC
* Lesion:
* Part 1: evaluable lesion (including skin or bone lesion only)
* Part 2: measurable lesion per RECIST v1.1
* Prior systemic Treatment
* Part 1: HR-positive/HER2-negative BC
* At least 1 line of SOC, including CDK4/6 inhibitor therapy and Endocrine Therapy, for advanced or metastatic disease.
* Prior chemotherapy in the metastatic setting is allowed.
* Part 1: HR-positive/HER2-positive BC
* At least 1 prior treatment of approved HER2 targeting therapy.
* Part 1: Solid Tumors other than BC
* Participants with no standard therapy available or for which no local regulatory approved standard therapy is available that would confer significant clinical benefit in the medical judgement of the investigator.
* Part 2A: At least 1 prior systemic therapy for advanced or metastatic disease, including CDK4/6 inhibitor treatment and ET.
* Parts 2B: At least 1 prior endocrine therapy for advanced or metastatic disease. Progression during treatment or within 12 months of completion of adjuvant endocrine therapy is acceptable.
* Part 2B: Up to 1 prior line of chemotherapy for advanced/metastatic disease is allowed.
* General Inclusion Criteria
* Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) 0 or 1
* Adequate renal, liver, and bone marrow function
* Resolved acute effects of any prior therapy to baseline severity

Exclusion Criteria:

* All Study Parts: Permanent treatment discontinuation from prior CDK 4 and/or CDK2 inhibitor due to treatment related toxicity.
* Part 2B and 1C: Prior treatment with any CDK 4/6 inhibitor, or SERDs (e.g. fulvestrant), or everolimus, or any agent whose mechanism of action is to inhibit the PI3K-mTOR pathway for advanced disease.
* Parts 2B and 2C: Prior treatment with any CDK4/6 inhibitor for advanced disease.
* Parts 2B and 2C: Prior treatment with an investigational endocrine therapy for advanced disease.
* Part 2C: Prior neoadjuvant or adjuvant treatment with a nonsteroidal aromatase inhibitor AI (ie, anastrozole or letrozole) with disease recurrence while on or within 12 months of completing treatment.
* Part 2C: Any prior systemic treatment for advanced disease.
* Prior irradiation to >25% of the bone marrow
* Current use of drugs which have a risk for QTc prolongation
* Current use or anticipated need for food or drugs that are known strong CYP3A4/5, strong UGT2B7 or UGT1A9 inhibitors or inducers
* Participation in other studies involving investigational drug(s) within 4 weeks prior to study entry

  * Participants with any other active malignancy within 3 years prior to enrollment except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the cervix, Bowen's disease
  * Major surgery within 4 weeks prior to study entry
  * Radiation therapy within 4 weeks prior to study entry.
  * Clinically important hypertension
  * Known or suspected hypersensitivity to PF-07220060, PF-07104091, letrozole, fulvestrant, or goserelin (or equivalent to induce chemical menopause if applicable)
* Known abnormalities in coagulation. Anticoagulation with subcutaneous heparin or prophylactic doses of anticoagulant are allowed
* Known active uncontrolled or symptomatic central nervous system (CNS) metastases
* Active inflammatory GI disease
* Current use or anticipated need for Proton Pump Inhibitors (PPI) within 14 days prior to first dose of the study intervention
* Previous high-dose chemotherapy requiring stem cell rescue
* Participants with active, uncontrolled bacterial, fungal, or viral infection, including hepatitis B virus (HBV), hepatitis C virus (HCV), and known human immunodeficiency virus (HIV) or acquired immunodeficiency syndrome (AIDS) related illness
* Other protocol specific exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2022-03-14 (Actual); Primary Completion 2026-08-23 (Estimated); Study Completion 2026-08-23 (Estimated)

PRIMARY OUTCOMES:
Dose Escalation: Number of participants with Dose-limiting toxicities (DLT) during first cycle | Cycle 1 (28 days)
  Number of participants with DLTs, which are typically Grade 3 or higher adverse events will be summarized by dose level
Number of participants with treatment emergent adverse events (AEs) | From baseline until end of study treatment or study completion (approximately 2 years)
Incidence of participants with clinical laboratory abnormalities | From baseline until end of study treatment or study completion (approximately 2 years)
Number of participants with vital signs abnormalities | From baseline until end of study treatment or study completion (approximately 2 years)
Number of participants with corrected QT (QTc) interval | From baseline until end of study treatment or study completion (approximately 2 years)
  Determine the effect of the drug on QT prolongation. The number and percentage of participants who experienced QT interval prolongation will be summarized by dose level

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) of PF-07220060 and PF-07104091 together after a single dose and multiple dose | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
Time to maximum plasma concentration (Tmax) of PF-07220060 and PF-07104091 together after a single dose and multiple dose | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
Area under the concentration versus time curve from time zero to the last quantifiable time point prior to the next dose (AUClast) of PF-07220060 and PF-07104091 together | Day 1 and Day 15 of Cycle 1 (each cycle is 28 days)
Objective response rate (ORR) of PF-07220060 and PF-07104091 together in dose escalation and together in combination with fulvestrant or letrozole | From baseline through disease progression or study completion (approximately 2 years)
  Percentage of participants with a best ORR of complete response (CR) or partial response (PR) using RECIST 1.
To evaluate the preliminary antitumor activity of PF-07220060 and PF-07104091 together in dose escalation and together in combination with fulvestrant or letrozole by time to event endpoints | From baseline through time to event on study or study completion (approximately 2 years)
  Time from first assessment of event endpoint to last assessment of using RECIST 1.1
Duration of Response (DoR) of PF-07220060 and PF-07104091 together in dose escalation and together in combination with fulvestrant or letrozole | From baseline through time to event on study or study completion (approximately 2 years)
  DoR is defined as the time from first documentation of CR or PR to date of first documentation of progressive disease/pharmacodynamic (PD) or death due to any cause, whichever occurs first
Progression-Free Survival (PFS) of PF-07220060 and PF-07104091 together in dose escalation and together in combination with fulvestrant or letrozole | From baseline through time to event on study or study completion (approximately 2 years)
  PFS is defined as time from start date of treatment to the date of first documentation of PD or death due to any cause
Time to Progression (TTP) of PF-07220060 and PF-07104091 together in dose escalation and together in combination with fulvestrant or letrozole | From baseline through time to event on study or study completion (approximately 2 years)
  TTP is defined as the time from start date of treatment to the date of the first documentation of PD

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (50):
- United States (11):
  - Administrative Address: UCLA Hematology/Oncology, Los Angeles, California
  - Ronald Reagan UCLA Medical Center, Los Angeles, California
  - UCLA Hematology/Oncology, Los Angeles, California
  - UCLA Hematology / Oncology-Parkside, Santa Monica, California
  - UCLA Hematology/Oncology-Santa Monica, Santa Monica, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - START Midwest, Grand Rapids, Michigan
  - Saint Luke's Cancer Institute, Kansas City, Missouri
  - Texas Oncology-Baylor Charles A. Sammons Cancer Center, Dallas, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Swedish Medical Center, Seattle, Washington
- Argentina (4):
  - Clinica Viedma S. A, Viedma, Río Negro Province
  - Centro Oncologico Korben, Buenos Aires
  - Clínica Universitaria Reina Fabiola, Córdoba
  - Fundación CORI para la Investigación y Prevención del Cáncer, La Rioja
- Brazil (5):
  - ONCOSITE - Centro de Pesquisa Clinica em Oncologia, Ijuí, Rio Grande do Sul
  - Centro Gaucho Integrado De Oncologia, Hematologia, Ensino E Pesquisa, Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisa Clínica - Área Administrativa, Porto Alegre, Rio Grande do Sul
  - Fundação Pio XII - Hospital de Câncer de Barretos, Barretos, São Paulo
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda, São Paulo
- Bulgaria (5):
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia, Sofia (stolitsa)
  - Specialized Hospital for Active Treatment of Oncology - Haskovo, Haskovo
  - Complex Oncology Center - Plovdiv EOOD, Plovdiv
  - Multiprofile Hospital for Active Treatment Serdika EOOD, Sofia
  - Complex Oncology Center - Vratsa, Vratsa
- China (7):
  - The First Hospital of Jilin University, Changchun, Jilin
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute & Hospital, Tianjin, Tianjin Municipality
  - Sir Run Run Shaw Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
- Czechia (3):
  - Fakultni nemocnice Olomouc, Olomouc, Olomoucký kraj
  - Fakultni nemocnice Bulovka, Prague, Praha 8
  - Vseobecna fakultni nemocnice v Praze, Prague
- Mexico (3):
  - Instituto Nacional de Cancerologia, Mexico City, Mexico City
  - Hospital Universitario "Dr. Jose Eleuterio Gonzalez", Monterrey, Nuevo León
  - Mérida Investigación Clínica, Mérida, Yucatán
- South Africa (6):
  - FARMOVS, Bloemfontein, Free State
  - 15 Eton Road, Johannesburg, Gauteng
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - WCR Office, Johannesburg, Gauteng
  - Wits Clinical Research, Johannesburg, Gauteng
  - Wilgers Oncology Centre, Pretoria, Gauteng
- Spain (6):
  - CHUS - Hospital Clinico Universitario, Santiago de Compostela, A Coruña [LA Coruña]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [barcelona]
  - Hospital Clínic de Barcelona, Barcelona, Catalunya [cataluña]
  - Hospital Universitario 12 de Octubre, Madrid, Madrid, Comunidad de
  - Hospital Universitario HM Sanchinarro, Madrid, Madrid, Comunidad de
  - Hospital Universitario Virgen Del Rocio, Seville

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4391002